CLINICAL TRIAL: NCT04103034
Title: A Single/Multiple Ascending Dose Phase 1 Study of the Safety, Tolerability and Pharmacologic Activity of BT200 in Normal Human Volunteers
Brief Title: A SAD/MAD Study of Safety, Tolerability and Pharmacologic Activity of BT200 in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Band Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BT200-01
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Cerebrovascular Stroke; Large-Artery Atherosclerosis (Embolus/Thrombosis); Intracranial Arteriosclerosis
Keywords: Secondary Stroke Prevention
MeSH Terms: conditions — Stroke; Embolism; Thrombosis; Intracranial Arteriosclerosis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- BT200 0.18mg (Experimental): Subjects will receive a single subcutaneous dose of BT200 0.18mg
  Interventions: Drug: BT200
- BT200 0.6mg (Experimental): Subjects will receive a single subcutaneous dose of BT200 0.6mg
  Interventions: Drug: BT200
- BT200 1.8mg (Experimental): Subjects will receive a single subcutaneous dose of BT200 1.8mg
  Interventions: Drug: BT200
- BT200 6.0mg (Experimental): Subjects will receive a single subcutaneous dose of BT200 6.0mg
  Interventions: Drug: BT200
- BT200 12.0mg (Experimental): Subjects will receive a single subcutaneous dose of BT200 12.0mg
  Interventions: Drug: BT200
- BT200 24.0mg (Experimental): Subjects will receive a single subcutaneous dose of BT200 24.0mg
  Interventions: Drug: BT200
- BT200 24.0mg rep (Experimental): Subjects will receive a single subcutaneous (SC) dose of BT200 24.0mg by gradual SC infusion
  Interventions: Drug: BT200
- Placebo SAD (Placebo Comparator): Subjects will receive a single subcutaneous dose of placebo
  Interventions: Drug: Placebo
- BT200 loading dose 12.0mg, maintenance doses of 12.0 mg (Experimental): Subjects will receive an initial subcutaneous loading doses of BT200 12.0mg followed by 4 weekly (every 7 days) maintenance doses of BT200 12.0mg
  Interventions: Drug: BT200
- BT200 loading doses 24.0mg, maintenance doses of 24.0 mg (Experimental): Subjects will receive an initial subcutaneous loading dose of BT200 24mg followed by 4 weekly (every 7 days) maintenance doses of BT200 24mg
  Interventions: Drug: BT200
- Placebo MAD (Placebo Comparator): Subjects will receive an initial subcutaneous loading dose of Placebo followed by 4 weekly (every 7 days) maintenance doses of placebo
  Interventions: Drug: Placebo
- BT200 48.0mg + desmopressin challenge (Experimental): Subjects will receive a single subcutaneous dose of BT200 48.0mg followed by IV infusion (over 30 min) of 0.3µg/kg desmopressin administered 24 hours after single dose of BT200
  Interventions: Drug: BT200; Drug: Desmopressin
- Placebo + desmopressin challenge dose (Placebo Comparator): Subjects will receive a single subcutaneous dose of placebo followed by IV infusion (over 30 min of 0.3µg/kg desmopressin administered 24 hours after single dose of placebo
  Interventions: Drug: BT200; Drug: Desmopressin
- Placebo infusion (Placebo Comparator): Subjects will receive a single IV dose of placebo administered over 24 hours
  Interventions: Drug: Placebo
- BT200 36.0mg (Experimental): Subjects will receive a single subcutaneous (SC) dose of BT200 36.0mg by gradual SC infusion
  Interventions: Drug: BT200
- BT200 48.0 mg (Experimental): Subjects will receive a single subcutaneous dose (SC) of BT200 48.0mg by gradual SC infusion
  Interventions: Drug: BT200
- BT200 18.0 mg (Experimental): Subjects will receive a single subcutaneous (SC) dose of BT200 18.0mg by gradual SC infusion
  Interventions: Drug: BT200
- BT200 24mg IV infusion (Experimental): Subjects will receive a single IV dose of BT200 24mg administered over 24 hours
  Interventions: Drug: BT200

INTERVENTIONS:
Drug: BT200 — BT200 is a PEGylated synthetic RNA oligonucleotide
  Arms: BT200 0.18mg; BT200 0.6mg; BT200 1.8mg; BT200 12.0mg; BT200 18.0 mg; BT200 24.0mg; BT200 24.0mg rep; BT200 24mg IV infusion; BT200 36.0mg; BT200 48.0 mg; BT200 48.0mg + desmopressin challenge; BT200 6.0mg; BT200 loading dose 12.0mg, maintenance doses of 12.0 mg; BT200 loading doses 24.0mg, maintenance doses of 24.0 mg; Placebo + desmopressin challenge dose
Drug: Desmopressin — Sterile solution for injection
  Other Names: MINIRIN® Injection
  Arms: BT200 48.0mg + desmopressin challenge; Placebo + desmopressin challenge dose
Drug: Placebo — Sterile saline for injection
  Arms: Placebo MAD; Placebo SAD; Placebo infusion

SUMMARY:
Study BT200-01 is a first in human (FIH) study in male and female normal human volunteers (NHVs) that uses an Integrated Protocol Design. This Phase 1 study will comprise 4 sub-parts: Part A, a single ascending dose (SAD) study; Part B, a multiple ascending dose (MAD) study; Part C, a desmopressin challenge study to explore (i) whether desmopressin could be used as an antidote, and/or (ii) whether desmopressin stimulated vonWillebrand Factor (VWF) release is overcome with increasing BT200 doses; and Part D, a relative bioavailability (BA) study.

The primary objective of this study is to assess the safety and tolerability profile of BT200 in NHVs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers, age ≥ 18 years old at screening
2. If female, must be post-menopausal or status post hysterectomy
3. Able to comprehend and to give informed consent
4. Able to cooperate with the Investigator, to comply with the requirements of the study, and to complete the full sequence of protocol-related procedures

Exclusion Criteria:

1. Clinically significant medical history (including von Willebrand Disease, thrombocytopathy, or any type of bleeding diathesis) or ongoing chronic illness that would jeopardize the safety of the subject or compromise the quality of the data derived from his/her participation in this study
2. Clinically relevant abnormal findings on physical examination or clinically relevant laboratory abnormalities
3. History of infusion hypersensitivity reactions, significant drug allergy, or anaphylactic reactions
4. Substance abuse, mental illness, or any reason that makes it unlikely in the judgment of the Investigator for the subject to be able to comply fully with study procedures
5. Use of medication during 2 weeks before the start of the study, which in the judgment of the Investigator may adversely affect the subject's welfare or the integrity of the study's results
6. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days or 5 elimination half-lives (whichever is longer) prior to treatment start

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Gilbert, MD, Study Director — Band Therapeutics; Ulla Derhaschnig, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Buchtele N, Schwameis M, Gilbert JC, Schorgenhofer C, Jilma B. Targeting von Willebrand Factor in Ischaemic Stroke: Focus on Clinical Evidence. Thromb Haemost. 2018 Jun;118(6):959-978. doi: 10.1055/s-0038-1648251. Epub 2018 May 30. PMID 29847840
- [Result] Kovacevic KD, Grafeneder J, Schorgenhofer C, Gelbenegger G, Gager G, Firbas C, Quehenberger P, Jilma-Stohlawetz P, Bileck A, Zhu S, Gilbert JC, Beliveau M, Jilma B, Derhaschnig U. The von Willebrand factor A-1 domain binding aptamer BT200 elevates plasma levels of von Willebrand factor and factor VIII: a first-in-human trial. Haematologica. 2022 Sep 1;107(9):2121-2132. doi: 10.3324/haematol.2021.279948. PMID 34818873
- [Result] Denis CV, Lenting PJ. How to keep the factor VIII/von Willebrand factor complex in the circulation. Haematologica. 2022 Sep 1;107(9):2011-2013. doi: 10.3324/haematol.2021.280222. No abstract available. PMID 34818875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Medical University of Vienna Phase 1 Unit's database of Normal Human Volunteers and a recruitment vendor was also employed.
Groups:
- BT200 Loading Dose 24.0mg, Maintenance Doses of 12.0 mg: Subjects will receive an initial subcutaneous loading doses of BT200 24.0mg followed by 4 weekly (every 7 days) maintenance doses of BT200 12.0mg
  BT200: BT200 is a PEGylated synthetic RNA oligonucleotide
- BT200 Loading Doses 48.0mg, Maintenance Doses of 24.0 mg: Subjects will receive an initial subcutaneous loading dose of BT200 48mg followed by 4 weekly (every 7 days) maintenance doses of BT200 24mg
  BT200: BT200 is a PEGylated synthetic RNA oligonucleotide
- BT200 18.0 mg: Subjects will receive a single subcutaneous dose of BT200 18.o mg
Period: Overall Study
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | Placebo SAD | BT200 Loading Dose 24.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 48.0mg, Maintenance Doses of 24.0 mg | Placebo MAD | BT200 48.0mg + Desmopressin Challenge | Placebo + Desmopressin Challenge Dose | Placebo Infusion | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT200 24mg IV Infusion
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 20 | 6 | 6 | 4 | 6 | 2 | 2 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 19 | 6 | 0 | 2 | 6 | 2 | 2 | 5 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- BT 200 24mg IV Infusion: Subjects will receive a single IV dose of BT200 24mg administered over 24 hours
- Total: Total of all reporting groups
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | Placebo SAD | BT200 Loading Dose 12.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 24.0mg, Maintenance Doses of 24.0 mg | Placebo MAD | BT200 48.0mg + Desmopressin Challenge | Placebo + Desmopressin Challenge Dose | Placebo Infusion | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT 200 24mg IV Infusion | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 20 | 6 | 6 | 4 | 6 | 2 | 2 | 6 | 6 | 6 | 6 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 19 | 6 | 5 | 4 | 6 | 2 | 2 | 6 | 6 | 6 | 6 | 109
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 11
  Male | 5 | 6 | 4 | 6 | 6 | 6 | 4 | 18 | 5 | 6 | 3 | 5 | 2 | 2 | 6 | 5 | 6 | 6 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 20 | 6 | 6 | 4 | 6 | 2 | 2 | 6 | 6 | 6 | 6 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 5 | 6 | 6 | 5 | 6 | 6 | 6 | 20 | 6 | 5 | 4 | 6 | 2 | 1 | 6 | 6 | 5 | 5 | 106
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 20 | 6 | 6 | 4 | 6 | 2 | 2 | 6 | 6 | 6 | 6 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Any AE or bleeding event related to study treatment
Time Frame: Baseline through 8 weeks after dosing up to 56 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | Placebo SAD | BT200 Loading Dose 12.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 24.0mg, Maintenance Doses of 24.0 mg | Placebo MAD | BT200 48.0mg + Desmopressin Challenge | Placebo + Desmopressin Challenge Dose | Placebo Infusion | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT200 24mg IV Infusion
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 20 | 6 | 6 | 4 | 6 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 4 | 3 | 3 | 3 | 0 | 0 | 0 | 3 | 2 | 0

2. Secondary Outcome: Measured Area Under the Curve (AUC)
Description: Measured Area Under the Curve at timepoints pre-dose, 0.5h, 1h, 4h, 8h,14h, 24h, 48h, 72h, 96h, 168h, 14d, 21d, 28d, 42d, 56d post dose
Time Frame: Baseline through 8 weeks after dosing up to 56 days
Population: Per protocol population-(h*ug/mL)
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | BT200 Loading Dose 24.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 48.0mg, Maintenance Doses of 24.0 mg | BT200 48.0mg + Desmopressin Challenge | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT200 24mg IV Infusion
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ug/mL | 1.159 (0.72594) | 5.405 (2.1113) | 11.50 (6.5663) | 64.39 (22.534) | 161.6 (43.427) | 259.5 (99.216) | 265.3 (59.127) | 409.4 (32.347) | 806.8 (187.25) | 675.9 (204.80) | 366.2 (78.610) | 638.8 (90.467) | 220.3 (64.58) | 555.4 (126.99)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma Concentration measured at pre-dose, 0.5h, 1h, 4h, 8h,14h, 24h, 48h, 72h, 96h, 168h, 14d, 21d, 28d, 42d, 56d
Time Frame: Baseline through 8 weeks after dosing up to 56 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | BT200 Loading Dose 24.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 48.0mg, Maintenance Doses of 24.0 mg | BT200 48.0mg + Desmopressin Challenge | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT200 24mg IV Infusion
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ug/mL | 0.01025 (0.0055459) | 0.04688 (0.018522) | 0.09432 (0.035964) | 0.5087 (0.18430) | 1.258 (0.35540) | 2.092 (0.07627) | 2.080 (0.46217) | 3.013 (0.25185) | 5.823 (1.3606) | 6.598 (2.6719) | 3.248 (11724) | 5.525 (0.95429) | 1.742 (0.49545) | 5.037 (1.3953)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum plasma concentration measured at pre-dose, 0.5h, 1h, 4h, 8h,14h, 24h, 48h, 72h, 96h, 168h, 14d, 21d, 28d, 42d, 56d
Time Frame: Baseline through 8 weeks after dosing up to 56 days
Population: per protocol population
Measure: Mean (Standard Deviation); unit: (h)
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | BT200 Loading Dose 24.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 48.0mg, Maintenance Doses of 24.0 mg | BT200 48.0mg + Desmopressin Challenge | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT200 24mg IV Infusion
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
(h) | 111.867 (111.7018) | 80.433 (20.2385) | 72.364 (22.0757) | 100.239 (53.4433) | 72.761 (21.4536) | 100.247 (38.5146) | 88.517 (19.7697) | 29.892 (25.8845) | 12.811 (17.9877) | 105.919 (18.9321) | 139.647 (46.6683) | 107.892 (113.4475) | 100.247 (38.5146) | 23.864 (0.2642)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of screening up to 56 days post dose
Arm/Group | BT200 0.18mg | BT200 0.6mg | BT200 1.8mg | BT200 6.0mg | BT200 12.0mg | BT200 24.0mg | BT200 24.0mg Rep | Placebo SAD | BT200 Loading Dose 12.0mg, Maintenance Doses of 12.0 mg | BT200 Loading Doses 24.0mg, Maintenance Doses of 24.0 mg | Placebo MAD | BT200 48.0mg + Desmopressin Challenge | Placebo + Desmopressin Challenge Dose | Placebo Infusion | BT200 36.0mg | BT200 48.0 mg | BT200 18.0 mg | BT200 24mg IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/20 | 0/6 | 0/6 | 0/4 | 0/6 | 0/2 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 1/20 | 0/6 | 1/6 | 0/4 | 0/6 | 0/2 | 0/2 | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6 | 4/6 | 4/6 | 5/6 | 6/6 | 5/6 | 16/20 | 6/6 | 6/6 | 4/4 | 5/6 | 1/2 | 1/2 | 4/6 | 4/6 | 5/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT200 0.18mg (N=6) | BT200 0.6mg (N=6) | BT200 1.8mg (N=6) | BT200 6.0mg (N=6) | BT200 12.0mg (N=6) | BT200 24.0mg (N=6) | BT200 24.0mg Rep (N=6) | Placebo SAD (N=20) | BT200 Loading Dose 12.0mg, Maintenance Doses of 12.0 mg (N=6) | BT200 Loading Doses 24.0mg, Maintenance Doses of 24.0 mg (N=6) | Placebo MAD (N=4) | BT200 48.0mg + Desmopressin Challenge (N=6) | Placebo + Desmopressin Challenge Dose (N=2) | Placebo Infusion (N=2) | BT200 36.0mg (N=6) | BT200 48.0 mg (N=6) | BT200 18.0 mg (N=6) | BT200 24mg IV Infusion (N=6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 3 SAE of back pain considered unrelated to study drug.
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 3 SAE of humerus fracture considered unrelated to study dug
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 3 SAE of intervertebral disc protrusion considered unrelated to study drug
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 3 SAE of prostate cancer considered unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT200 0.18mg (N=6) | BT200 0.6mg (N=6) | BT200 1.8mg (N=6) | BT200 6.0mg (N=6) | BT200 12.0mg (N=6) | BT200 24.0mg (N=6) | BT200 24.0mg Rep (N=6) | Placebo SAD (N=20) | BT200 Loading Dose 12.0mg, Maintenance Doses of 12.0 mg (N=6) | BT200 Loading Doses 24.0mg, Maintenance Doses of 24.0 mg (N=6) | Placebo MAD (N=4) | BT200 48.0mg + Desmopressin Challenge (N=6) | Placebo + Desmopressin Challenge Dose (N=2) | Placebo Infusion (N=2) | BT200 36.0mg (N=6) | BT200 48.0 mg (N=6) | BT200 18.0 mg (N=6) | BT200 24mg IV Infusion (N=6)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Root canal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (6) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 6 (7) | 4 (10) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain uppe (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gammaglutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parasthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04103034/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT04103034/SAP_001.pdf